CLINICAL TRIAL: NCT01689233
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 18-Month Safety and Efficacy Study of TRx0237 in Subjects With Mild Alzheimer's Disease
Brief Title: Safety and Efficacy Study Evaluating TRx0237 in Subjects With Mild Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRx-237-005
Record Dates: First submitted 2012-09-14; First posted 2012-09-21 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer Disease; TRx0237; AD; Neurodegenerative Diseases; Dementia; Brain Diseases
MeSH Terms: conditions — Alzheimer Disease; Neurodegenerative Diseases; Dementia; Brain Diseases | interventions — hydromethylthionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRx0237 200 mg/day (Experimental)
  Interventions: Drug: TRx0237 200 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRx0237 200 mg/day — TRx0237 100 mg tablets will be administered twice daily.
  Arms: TRx0237 200 mg/day
Drug: Placebo — Placebo tablets will be administered twice daily. The active placebo tablets include 4 mg of TRx0237 as a urinary and fecal colorant to maintain blinding; hence the placebo group will receive a total of 8 mg/day of TRx0237.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of TRx0237 in the treatment of subjects with mild Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of all cause dementia and probable Alzheimer's disease
* Clinical Dementia Rating (CDR) total score of 0.5 or 1 (mild) and MMSE score of 20-26 (inclusive)
* Age <90 years
* Modified Hachinski ischemic score of ≤4
* Females, if of child-bearing potential, must practice true abstinence or be competent to use adequate contraception and agree to maintain this throughout the study
* Subject, and/or, in the case of reduced decision-making capacity, legally acceptable representative(s) consistent with national law is/are able to read, understand, and provide written informed consent
* Has one (or more) identified adult caregiver who is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; either lives with the subject or sees the subject for ≥2 hours/day ≥3 days/week; agrees to accompany the subject to each study visit; and is able to verify daily compliance with study drug
* If currently taking an acetylcholinesterase inhibitor and/or memantine at the time of Screening, the subject must have been taking such medication(s) for ≥3 months. The dosage regimen must have remained stable for ≥6 weeks and it must be planned to remain stable throughout participation in the study.
* Able to comply with the study procedures

Exclusion Criteria:

* Significant central nervous system (CNS) disorder other than Alzheimer's disease
* Significant focal or vascular intracranial pathology seen on brain MRI scan
* Clinical evidence or history of stroke, transient ischemic attack, significant head injury or other unexplained or recurrent loss of consciousness ≥15 minutes
* Epilepsy
* Major depressive disorder, schizophrenia, or other psychotic disorders, bipolar disorder, substance (including alcohol) related disorders
* Metal implants in the head (except dental), pacemaker, cochlear implants, or any other non-removable items that are contraindications to MRI
* Resides in hospital or moderate to high dependency continuous care facility
* History of swallowing difficulties
* Pregnant or breastfeeding
* Glucose-6-phosphate dehydrogenase deficiency
* History of significant hematological abnormality or current acute or chronic clinically significant abnormality
* Abnormal serum chemistry laboratory value at Screening deemed to be clinically relevant by the investigator
* Clinically significant cardiovascular disease or abnormal assessments
* Preexisting or current signs or symptoms of respiratory failure
* Concurrent acute or chronic clinically significant immunologic, hepatic, or endocrine disease (not adequately treated) and/or other unstable or major disease other than Alzheimer's disease
* Diagnosis of cancer within the past 2 years prior to Baseline (other than basal cell or squamous cell skin cancer or Stage 1 prostate cancer) unless treatment has resulted in complete freedom from disease for at least 2 years
* Prior intolerance or hypersensitivity to methylthioninium-containing drug, similar organic dyes, or any of the excipients
* Treatment currently or within 3 months before Baseline with any of the following medications (unless otherwise noted):

  * Tacrine
  * Clozapine, olanzapine (and there is no intent to initiate therapy during the course of the study)
  * Carbamazepine, primidone
  * Drugs with a warning or precaution in the labeling of methemoglobinemia at approved doses
* Current or prior participation in a clinical trial as follows:

  * Clinical trial of a product for cognition in which the last dose was received within 90 days prior to Screening (unless confirmed to have been randomized to placebo)
  * A clinical trial of a drug, biologic, device, or medical food in which the last dose/administration was received within 28 days prior to Baseline

Max Age: 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-cog11) | 78 weeks
Change from Baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23) | 78 weeks
Number of study participants who tolerate oral doses of TRx0237 as determined by safety parameter changes | 78 weeks
  Safety parameters include adverse events, vital signs, methemoglobin and oxygen saturation, physical and neurological examinations, laboratory tests (hematology, serum chemistry, and urinalysis), electrocardiograms, potential for serotonin toxicity, brain magnetic resonance imaging (MRI), and potential for suicide or self-harm.

SECONDARY OUTCOMES:
Change from Baseline in Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | 78 weeks
Change from Baseline in Mini-Mental Status Examination (MMSE) | 78 weeks
Change from Baseline in Neuropsychiatric Inventory (NPI) | 78 weeks
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | 78 weeks
Change in expected decline of whole brain volume as measured by brain MRI | 78 weeks

OTHER OUTCOMES:
Change in resource utilization using the Resource Utilization in Dementia (RUD) Lite | 78 weeks
Change in cerebrospinal fluid biomarkers of Alzheimer's Disease in subjects who separately consent to lumbar puncture | 78 weeks
Compare the influence of Apolipoprotein E genotype on the primary and selected secondary outcomes in subjects by or for whom legally acceptable consent is separately provided | 78 weeks
Reduction in glucose uptake decline in the temporal lobe on 18F-fluorodeoxyglucose positron emission tomography (FDG-PET) imaging | 78 weeks
Change in expected increase in ventricular volume as measured by brain MRI | 78 weeks
Change in expected decline in hippocampal volume as measured by brain MRI | 78 weeks

CONTACTS AND LOCATIONS:
Locations (95):
- United States (58):
  - Xenoscience, Inc / 21st Century Neurology, Phoenix, Arizona
  - NoesisPharma Clinical Trials, Phoenix, Arizona
  - CITrials, Bellflower, California
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Southern California Research, LLC, Fountain Valley, California
  - Feldman, Robert MD, Laguna Hills, California
  - Synergy East, Lemon Grove, California
  - Collaborative Neuroscience Network, Long Beach, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - Anderson Clinical Research, Redlands, California
  - Pacific Research Network, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Neurological Research Institute, Santa Monica, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Mile High Research Center, Denver, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Coastal Connecticut Research, LLC, New London, Connecticut
  - Research Center for Clinical Studies, Inc, Norwalk, Connecticut
  - JEM Research, Atlantis, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Compass Research, LLC, Orlando, Florida
  - The Roskamp Institute, Inc., Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Compass Research, LLC - North Clinic, The Villages, Florida
  - Premiere Research Institute (Palm Beach Neurology), West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Neurostudies.net, Decatur, Georgia
  - Alexian Brothers Neurosciences Institute, Elk Grove, Illinois
  - Ruan Neurology Clinic and Research Center, Des Moines, Iowa
  - CBH Health, LLC, Rockville, Maryland
  - Quest Research Institute, Farmington Hills, Michigan
  - Neurological Research Center - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Olive Branch Family Medical, Olive Branch, Mississippi
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - Memory Enhancement Centers of America, Inc, Eatontown, New Jersey
  - Advanced Memory Research Institute of NJ PC, Toms River, New Jersey
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - Neurological Associates of Albany, P. C., Albany, New York
  - MedicalPsych Care, PLLC, Elmsford, New York
  - Columbia University Taub Institute, New York, New York
  - Research Foundation for Mental Hygiene, Inc., Orangeburg, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Clinical Trials of America, Inc, Winston-Salem, North Carolina
  - Neurobehavorial Clinical Research, Canton, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - RI Hospital, Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Clinical Neuroscience Solutions CNS Healthcare, Memphis, Tennessee
  - Senior Adults Specialty Research, Inc., Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - PRA Health Sciences, Salt Lake City, Utah
  - Independent Psychiatric Consultants, Waukesha, Wisconsin
- Discipline of Psychiatry, University of Queensland, Herston, Queensland, Australia
- Belgium (5):
  - University Hospital Brussels Department of Neurology, Brussels
  - University Hospital Gent Department of Neurology, Ghent
  - Jessa Hospital, Hasselt
  - Regional Hospital Sint-Trudo, Sint-Truiden
  - GasthuisZusters Antwerpen Sint-Augustinus, Wilrijk
- Canada (4):
  - University of British Columbia Hospital, Clinic for Alzheimer Disease and Related Disorders, Vancouver, British Columbia
  - Parkwood Institute, London, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Croatia (2):
  - University Hospital Centre Zagreb, Department of Neurology, Zagreb
  - University Psychiatric Hospital Vrapče, Zagreb
- Finland (2):
  - University of Eastern Finland, Brain Research Unit Mediteknia, Kuopio
  - Clinical Research Services Turku (CRST), Turku
- France (3):
  - Hôpitaux Civils de Colmar, Colmar
  - Hôpital La Grave, Toulouse
  - Hôpital de Charpennes, Villeurbanne
- Germany (5):
  - Neurozentrum Achim Dr. med. Andreas Mahler, Achim
  - University Medicine Berlin - Charité, CBF, Neurology, Berlin
  - Memory Clinic, ECRC, Berlin
  - Arzeneimittelforschung Leipzig GmbH, Leipzig
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie Zentrum für Nervenheilkunde - Universitätsklinikum Rostock, Rostock
- Italy (5):
  - A.O.U. Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
  - IRCCS San Giovanni di Dio - Fatebenefratelli, Brescia
  - Fondazione Universita 'G. D'Annunzio di Chieti, Chieti Scalo
  - Clinical Neurology Department of Neuroscience (DINOGMI) - University of Genoa, Genova
  - Azienda Ospedaliera Universitaria Sant'Andrea di Roma - Unita' di Neurologia, Roma
- Alzheimer Center Southwest Netherlands, Erasmus MC, Rotterdam, Netherlands
- Spain (4):
  - Fundacio ACE, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari Mútua de Terrassa, Terrassa
- United Kingdom (5):
  - Grampian NHS, Royal Cornhill Hospital, Aberdeen
  - Sussex Partnership NHS Foundation Trust, Cognitive Treatment and Research Unit, Crowborough
  - Re:Cogniton Health, London
  - Memory Assessment and Research Centre (MARC), Southampton
  - Kingshill Research Centre, Victoria Hospital, Swindon

REFERENCES:
- See also: Alzheimer's Survey — http://www.AlzheimersStudies.com